CLINICAL TRIAL: NCT03050619
Title: Characteristics of Patients Initiating Empagliflozin or Other Non-insulin Glucose Lowering Drugs in the United Kingdom
Brief Title: Characteristics of Empagliflozin Initiators
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245.122
Record Dates: First submitted 2016-08-25; First posted 2017-02-13 (Actual); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- New users of Empagliflozin: New users of empagliflozin
  Interventions: Drug: Empagliflozin
- New users of Other SGLT2 inhibitors: New users of other SGLT2 inhibitors
  Interventions: Drug: Other SGLT2 inhibitors
- New users of Other non-insulin GLDs: New users of other non-insulin GLDs
  Interventions: Drug: Other non-insulin GLDs

INTERVENTIONS:
Drug: Empagliflozin
  Groups: New users of Empagliflozin
Drug: Other SGLT2 inhibitors
  Groups: New users of Other SGLT2 inhibitors
Drug: Other non-insulin GLDs — metformin, sulfonylureas, DPP-4 inhibitors, GLP-1 agonists
  Groups: New users of Other non-insulin GLDs

SUMMARY:
Empagliflozin, a sodium glucose cotransporter 2 (SGLT-2) inhibitor, was launched in the United Kingdom (UK) in August 2014. It can be expected that patients initiating empagliflozin may differ in their characteristics from patients initiating other glucose lowering drugs (GLDs) that have been on the market longer (e.g. patients may have poorer glucose control). Therefore, the proposed study aims to characterize patients with T2DM in the UK initiating empagliflozin in terms of baseline characteristics, concomitant medications, and comorbidities compared to patients with type 2 diabetes mellitus (T2DM) initiating other SGLT-2 inhibitors or other non-insulin GLDs. Due to the mode of action, some patients taking empagliflozin have experienced weight loss in clinical trials. A theoretical possibility exists that empagliflozin may be used by patients without T2DM. Therefore, this study also aims to assess the potential off-label use of empagliflozin compared to other non-insulin GLDs.

DETAILED DESCRIPTION:
Study Design:

cross sectional

ELIGIBILITY:
Inclusion criteria:

All patients will be required to meet all of the following criteria:

* At least 12 months of continuous registration prior to the index date in a practice contributing up to standard (UTS) data to the Clinical Practice Research Datalink (CPRD). Infants younger than 1 year will not be required to have 12 months of continuous UTS registration in the CPRD.
* A new user of one of the index prescriptions (empagliflozin, other SGLT2 inhibitor, or non-insulin GLDs) or a fixed dose combination (FDC) with metformin.

Exclusion criteria:

There is no exclusion criterion in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: New users of empagliflozin and other non-insulin GLDs in the UK CPRD between 1 Aug 2014 to 1 Sep 2015
Sampling Method: Non-Probability Sample
Enrollment: 31908 (Actual)
Dates: Start 2016-09-10 (Actual); Primary Completion 2016-10-14 (Actual); Study Completion 2016-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Boehringer Ingelheim Investigational Site, Ingelheim, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All study participants had at least 12 months of continuous registration in the United Kingdom (UK) Clinical Practice Research Datalink (CPRD) prior to the study initiation which is a data source comprising primary care electronic medical record (EMR).
Groups:
- Empagliflozin: Subjects who initiated treatment with empagliflozin in the United Kingdom (UK) between 01 August 2014 and 01 September 2015.
- Other SGLT-2i: Subjects who initiated treatment with other sodium glucose cotransporter 2 inhibitors (SGLT-2i) in the UK between 01 August 2014 and 01 September 2015.
- Dipeptidyl Peptidase-4 Inhibitors (DPP-4i): Subjects who initiated treatment with DPP-4i in the UK between 01 August 2014 and 01 September 2015.
- Metformin: Subjects who initiated treatment with metformin in the UK between 01 August 2014 and 01 September 2015.
- Sulfonylureas (SU): Subjects who initiated treatment with SU in the UK between 01 August 2014 and 01 September 2015.
- Glucagon-like Peptide-1 (GLP-1) Agonists: Subjects who initiated treatment with GLP-1 agonists in the UK between 01 August 2014 and 01 September 2015.
Period: Overall Study
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Started | 129 | 3926 | 6416 | 14007 | 6079 | 1351
Completed | 129 | 3926 | 6416 | 14007 | 6079 | 1351
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients (older than 18 years), with a recorded type 2 diabetes mellitus (T2DM), who initiated treatment with empagliflozin, other SGLT-2i, or other commonly used non-insulin glucose lowering drugs (GLDs) (comprising DPP-4i, metformin, SU and GLP-1 agonists) between 01 August 2014 and 01 September 2015 were included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists | Total
Number analyzed (Participants) | 110 | 3407 | 5615 | 10370 | 5271 | 1155 | 25928
Age, Customized [Count of Participants; unit: Participants]
  18 - 35 years | 6 | 60 | 81 | 314 | 141 | 37 | 639
  36 - 49 years | 25 | 637 | 643 | 1748 | 753 | 224 | 4030
  50 - 64 years | 47 | 1683 | 1952 | 3858 | 1925 | 560 | 10025
  65 - 74 years | 22 | 862 | 1601 | 2576 | 1347 | 266 | 6674
  75 years and above | 10 | 165 | 1338 | 1874 | 1105 | 68 | 4560
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 1404 | 2406 | 4464 | 2284 | 571 | 11180
  Male | 59 | 2003 | 3209 | 5906 | 2987 | 584 | 14748

OUTCOME MEASURES:

1. Primary Outcome: Baseline Characteristics of Adults (as Measured by Demographics) With a Recorded Diagnosis of T2DM Starting Index Prescriptions in the UK
Description: Baseline characteristics of adults (as measured by demographics) with a recorded diagnosis of T2DM who initiated index prescriptions (empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists)) are presented.
Time Frame: Baseline
Population: All patients (older than 18 years), with a recorded T2DM, who initiated treatment with empagliflozin, other SGLT-2i, or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists) between 01 August 2014 and 01 September 2015 were included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Number analyzed (Participants) | 110 | 3407 | 5615 | 10370 | 5271 | 1155
Percentage of Participants
  Age (18 - 35 years) | 5.45 | 1.76 | 1.44 | 3.03 | 2.68 | 3.20
  Age (36 - 49 years) | 22.73 | 18.70 | 11.45 | 16.86 | 14.29 | 19.39
  Age (50 - 64 years) | 42.73 | 49.40 | 34.76 | 37.20 | 36.52 | 48.48
  Age (65 - 74 years) | 20.00 | 25.30 | 28.51 | 24.84 | 25.55 | 23.03
  Age (75 years and above) | 9.09 | 4.84 | 23.83 | 18.07 | 20.96 | 5.89
  Gender (Female) | 46.36 | 41.21 | 42.85 | 43.05 | 43.33 | 49.44
  Gender (Male) | 53.64 | 58.79 | 57.15 | 56.95 | 56.67 | 50.56

2. Primary Outcome: Baseline Characteristics of Adults (as Measured by Life Style Factors (Smoking and Alcohol Use)) With a Recorded Diagnosis of T2DM Starting Index Prescriptions in the UK
Description: Baseline characteristics of adults (as measured by life style factors (smoking and alcohol use)) with a recorded diagnosis of T2DM who initiated index prescriptions (empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists)) are presented. NA= NR (Not Reported) (variables for which patient counts were <5)
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Number analyzed (Participants) | 110 | 3407 | 5615 | 10370 | 5271 | 1155
Percentage of Participants
  Smoking (smoker) | 22.73 | 18.08 | 18.24 | 20.67 | 20.17 | 18.53
  Smoking (non-smoker) | 19.09 | 29.03 | 27.96 | 30.95 | 27.98 | 27.01
  Smoking (ex-smoker) | 58.18 | 52.89 | 53.80 | 48.20 | 51.79 | 54.46
  Smoking (Unknown) | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 0.18 | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality.
  Alcohol consumption (drinker) | 60.00 | 68.59 | 66.25 | 68.14 | 65.81 | 65.45
  Alcohol consumption (non-drinker) | 15.45 | 9.25 | 10.37 | 10.15 | 10.15 | 9.18
  Alcohol consumption (ex-drinker) | 22.73 | 19.81 | 21.25 | 17.04 | 20.32 | 23.03
  Alcohol consumption (Unknown) | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 2.35 | 2.14 | 4.67 | 3.72 | 2.34

3. Primary Outcome: Baseline Characteristics of Adults (as Measured by Life Style Factors (BMI)) With a Recorded Diagnosis of T2DM Starting Index Prescriptions in the UK
Description: Baseline characteristics of adults (as measured by life style factors (BMI)) with a recorded diagnosis of T2DM who initiated index prescriptions (empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists)) is presented. Mean and standard deviation (SD) of body mass index (BMI) measured is presented along with number of subjects with available data.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kilogram per square meter (kg/m2)
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Number analyzed (Participants) | 107 | 3357 | 5460 | 8964 | 4957 | 1133
Kilogram per square meter (kg/m2) | 35.43 (5.83) | 35.24 (6.82) | 32.13 (6.45) | 32.99 (6.83) | 31.61 (6.57) | 37.68 (6.72)

4. Primary Outcome: Baseline Characteristics of Adults (as Measured by Life Style Factors (Blood Pressure)) With a Recorded Diagnosis of T2DM Starting Index Prescriptions in the UK
Description: Baseline characteristics of adults (as measured by life style factors (blood pressure)) with a recorded diagnosis of T2DM who initiated index prescriptions (empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists)) is presented. Mean and standard deviation (SD) of Systolic blood pressure (SBP) and Diastolic blood pressure (DBP) measured is presented along with number of subjects with available data.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Number analyzed (Participants) | 110 | 3407 | 5615 | 10370 | 5271 | 1155
Millimeter of mercury (mmHg)
  SBP: number analyzed (Participants) | 106 | 3110 | 5173 | 8636 | 4722 | 1069
  SBP | 130.75 (14.72) | 133.52 (13.70) | 133.45 (14.61) | 135.02 (15.57) | 132.72 (14.86) | 133.84 (14.31)
  DBP: number analyzed (Participants) | 106 | 3121 | 5180 | 8649 | 4725 | 1068
  DBP | 77.02 (8.24) | 77.85 (8.91) | 76.02 (9.46) | 78.48 (10.19) | 76.78 (9.54) | 77.82 (8.67)

5. Primary Outcome: Baseline Characteristics of Adults (as Measured by Glycated Haemoglobin (HbA1c)) With a Recorded Diagnosis of T2DM Starting Index Prescriptions in the UK
Description: Baseline characteristics of adults (as measured by glycated haemoglobin (HbA1c)) with a recorded diagnosis of T2DM who initiated index prescriptions (empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists)) is presented. Mean and standard deviation (SD) of glycated haemoglobin (HbA1c) measured is presented along with number of subjects with available data.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimole per mole (mmol/mol)
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Number analyzed (Participants) | 97 | 2954 | 4849 | 8132 | 4290 | 1036
Millimole per mole (mmol/mol) | 77.34 (16.02) | 79.52 (17.62) | 73.83 (17.81) | 70.35 (20.98) | 78.05 (21.39) | 80.68 (18.07)

6. Primary Outcome: Baseline Characteristics of Adults (as Measured by Laboratory Tests) With a Recorded Diagnosis of T2DM Starting Index Prescriptions in the UK
Description: Baseline characteristics of adults (as measured by laboratory tests) with a recorded diagnosis of T2DM who initiated index prescriptions (empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists)) are presented. Mean and standard deviation (SD) of total cholesterol (TC), high-density lipoproteins level (HDL), Low-density lipoprotein level (LDL) and triglyceride level (TG) measured are presented along with number of subjects with available data.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimole per liter (mmol/L)
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Number analyzed (Participants) | 110 | 3407 | 5615 | 10370 | 5271 | 1155
Millimole per liter (mmol/L)
  TC: number analyzed (Participants) | 105 | 3256 | 5277 | 8978 | 4765 | 1066
  TC | 4.22 (1.00) | 4.33 (1.10) | 4.29 (1.09) | 4.89 (1.26) | 4.53 (1.27) | 4.37 (1.05)
  HDL: number analyzed (Participants) | 95 | 2993 | 4873 | 8319 | 4337 | 974
  HDL | 1.10 (0.25) | 1.13 (0.30) | 1.17 (0.33) | 1.19 (0.33) | 1.18 (0.35) | 1.10 (0.27)
  LDL: number analyzed (Participants) | 72 | 2423 | 3871 | 6484 | 3209 | 705
  LDL | 2.17 (0.85) | 2.19 (0.86) | 2.19 (0.90) | 2.70 (1.01) | 2.32 (0.97) | 2.22 (0.88)
  TG: number analyzed (Participants) | 75 | 2709 | 4332 | 7312 | 3699 | 848
  TG | 2.22 (1.33) | 2.38 (1.89) | 2.23 (1.63) | 2.34 (1.90) | 2.43 (1.99) | 2.50 (1.72)

7. Primary Outcome: Baseline Characteristics of Adults (as Measured by Estimated Glomerular Filtration Rate (eGFR)) With a Recorded Diagnosis of T2DM Starting Index Prescriptions in the UK
Description: Baseline characteristics of adults (as measured by estimated glomerular filtration rate (eGFR)) with a recorded diagnosis of T2DM who initiated index prescriptions (empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists)) is presented. Mean and standard deviation (SD) of estimated glomerular filtration rate (eGFR) measured is presented along with number of subjects with available data.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliliters per minute (ml/min)
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Number analyzed (Participants) | 107 | 3315 | 5467 | 9609 | 5020 | 1097
Milliliters per minute (ml/min) | 95.46 (16.94) | 93.42 (30.95) | 80.68 (24.65) | 87.64 (19.56) | 84.95 (23.12) | 90.27 (20.44)

8. Primary Outcome: Baseline Characteristics of Adults (as Measured by Creatinine Serum (SCR)) With a Recorded Diagnosis of T2DM Starting Index Prescriptions in the UK
Description: Baseline characteristics of adults (as measured by by creatinine serum (SCR)) with a recorded diagnosis of T2DM who initiated index prescriptions (empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists)) is presented. Mean and standard deviation (SD) of creatinine serum (SCR) measured is presented along with number of subjects with available data.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Number analyzed (Participants) | 107 | 3315 | 5467 | 9609 | 5020 | 1097
Micromoles per liter (umol/L) | 72.16 (16.62) | 74.52 (17.18) | 88.46 (38.30) | 78.46 (20.00) | 83.10 (33.18) | 77.16 (23.97)

9. Primary Outcome: Baseline Characteristics of Adults (as Measured by Comorbidities) With a Recorded Diagnosis of T2DM Starting Index Prescriptions in the UK
Description: Baseline characteristics of adults (as measured by comorbidities) with a recorded diagnosis of T2DM who initiated index prescriptions (empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists)) are presented.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Number analyzed (Participants) | 110 | 3407 | 5615 | 10370 | 5271 | 1155
Percentage of Participants
  Diabetes complications | 34.55 | 34.14 | 33.62 | 13.11 | 24.36 | 34.81
  Thyroid disorders | 8.18 | 9.30 | 9.39 | 8.52 | 8.97 | 11.00
  Cancer | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 4.05 | 7.25 | 5.97 | 7.95 | 4.59
  Cardiovascular disorders | 56.36 | 56.88 | 62.60 | 54.85 | 59.70 | 59.83
  Infections | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 2.03 | 3.69 | 2.64 | 3.68 | 3.64
  Kidney disease | 11.82 | 9.48 | 22.81 | 12.40 | 17.40 | 14.98
  Polycystic Ovary Syndrome (PCO), females only | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 1.78 | 1.37 | 1.52 | 1.80 | 3.33
  Obesity | 40.00 | 39.01 | 26.79 | 20.69 | 24.45 | 45.71
  Respiratory | 22.73 | 21.10 | 19.89 | 19.59 | 20.13 | 21.90
  Pancreatitis | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 1.14 | 0.89 | 1.02 | 1.37 | 0.52
  Bone disorders | 8.18 | 11.39 | 12.80 | 12.10 | 13.15 | 12.55

10. Primary Outcome: Baseline Characteristics of Adults (as Measured by Concomitant Medications) With a Recorded Diagnosis of T2DM Starting Index Prescriptions in the UK
Description: Baseline characteristics of adults (as measured by concomitant medications) with a recorded diagnosis of T2DM who initiated index prescriptions (empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists)) are presented. Subjects taking medication up to 60 days before index date are presented.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Number analyzed (Participants) | 110 | 3407 | 5615 | 10370 | 5271 | 1155
Percentage of Participants
  Insulin | 15.45 | 17.64 | 5.95 | 2.34 | 2.26 | 18.18
  Non-insulin GLDs | 96.36 | 95.42 | 89.26 | 10.49 | 78.54 | 92.81
  Cardiovascular medications | 70.91 | 74.76 | 76.31 | 60.35 | 69.42 | 77.40
  Lipid-regulating Drugs | 79.09 | 76.20 | 74.37 | 47.92 | 64.81 | 75.67
  Oral Corticosteroids | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 2.76 | 4.49 | 4.99 | 5.86 | 2.94
  Non-steroidal anti-inflammatory drugs | 8.18 | 10.92 | 8.39 | 9.47 | 8.06 | 11.69
  Psycholeptics | 5.45 | 5.14 | 5.40 | 5.73 | 6.00 | 6.49
  Antipsychotics | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 3.08 | 3.51 | 3.85 | 3.74 | 3.90
  Antidepressants | 31.82 | 26.71 | 22.87 | 21.41 | 23.20 | 33.94
  Opiates | 22.73 | 21.19 | 20.11 | 18.57 | 20.05 | 24.33
  Anti-Epilepsy, Anticonvulsants | 9.09 | 9.01 | 9.58 | 8.39 | 8.95 | 13.25
  Anti-Parkinson, Dopamine agonists | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 2.26 | 2.49 | 2.80 | 2.79 | 2.86
  Agents for dementia | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 0.18 | 0.80 | 0.58 | 0.61 | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality.

11. Secondary Outcome: Extent of Off-label Use
Description: To assess off-label use the number of study participants without a recorded diagnosis of T2DM was calculated for each exposure category (people with other types of diabetes, people without diabetes, people younger than 18 years old, and women during pregnancy and breastfeeding). For the assessment of drug use during the pregnancy and breastfeeding period, the look-back period was 270 days (9 months) before and including the index date. To assess the use in pediatric population, the study participants were stratified by age into adults (≥18 years of age) and pediatrics (<18 years of age).
Time Frame: Baseline
Population: All patients (without any age restriction), with or without a recorded diagnosis of diabetes, who initiated treatment with empagliflozin, other SGLT-2i, or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists) between 01 August 2014 and 01 September 2015 were included.
Measure: Number; unit: Participants
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Number analyzed (Participants) | 129 | 3926 | 6416 | 14007 | 6079 | 1351
Participants
  Gestational diabetes, pregnancy, or breastfeeding | 0 | 4 | 2 | 581 | 8 | 0
  Without any diabetes mellitus (DM) code | 0 | 3 | 13 | 1601 | 136 | 1
  Type 1 diabetes mellitus (T1DM) | 1 | 45 | 21 | 159 | 30 | 10
  Unspecified DM | 14 | 345 | 569 | 1054 | 478 | 122
  Other diabetes | 0 | 2 | 3 | 20 | 22 | 1
  Mixed codes of DM | 4 | 120 | 192 | 218 | 133 | 62
  Younger than 18 years with T2DM | 0 | 0 | 0 | 4 | 1 | 0

12. Secondary Outcome: Baseline Characteristics (as Measured by Demographics) of Patients Starting Index Prescriptions Off-label
Description: Baseline characteristics of patients (as measured by demographics) who initiated index prescriptions (empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists)) off-label are presented. Use of empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs in other types of diabetes (other than T2DM) or without diabetes or in people younger than 18 years old or in women during pregnancy or during breastfeeding is considered as off-label. As per CPRD guideline, no cell that contains <5 events should be reported to protect patient confidentiality. Since empagliflozin group reported <5 events for all off-label categories except for unspecified DM therefore baseline characteristics are presented for only unspecified DM category.
Time Frame: Baseline
Population: All patients older than 18 years with unspecified DM who initiated treatment with empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists) between 01 August 2014 and 01 September 2015 were included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Number analyzed (Participants) | 14 | 346 | 569 | 1049 | 478 | 122
Percentage of Participants
  Age (18 - 35 years) | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 2.60 | 0.88 | 11.44 | 2.51 | 4.10
  Age (36 - 49 years) | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 19.65 | 10.72 | 19.64 | 12.34 | 17.21
  Age (50 - 64 years) | 42.86 | 45.95 | 30.93 | 31.65 | 35.36 | 45.90
  Age (65 - 74 years) | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 24.86 | 30.23 | 21.64 | 25.10 | 25.41
  Age (75 years and above) | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 6.94 | 27.24 | 15.63 | 24.69 | 7.38
  Gender (Female) | 35.71 | 42.49 | 40.60 | 48.90 | 44.56 | 55.74
  Gender (Male) | 64.29 | 57.51 | 59.40 | 51.10 | 55.44 | 44.26

13. Secondary Outcome: Baseline Characteristics (as Measured by Life Style Factors (Smoking and Alcohol Use)) of Patients Starting Index Prescriptions Off-label
Description: Baseline characteristics of patients (as measured by life style factors (smoking and alcohol use)) who initiated index prescriptions (empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists)) off-label are presented. Use of empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs in other types of diabetes (other than T2DM) or without diabetes or in people younger than 18 years old or in women during pregnancy or during breastfeeding is considered as off-label. As per CPRD guideline, no cell that contains <5 events should be reported to protect patient confidentiality. Since empagliflozin group reported <5 events for all off-label categories except for unspecified DM therefore baseline characteristics are presented for only unspecified DM category. NA= NR (Not Reported) (variables for which patient counts were <5)
Time Frame: Baseline
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Number analyzed (Participants) | 14 | 346 | 569 | 1049 | 478 | 122
Percentage of Participants
  Smoking (smoker) | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 23.99 | 16.34 | 22.21 | 22.59 | 13.93
  Smoking (non-smoker) | 42.86 | 32.37 | 31.81 | 35.46 | 33.89 | 37.70
  Smoking (ex-smoker) | 35.71 | 43.64 | 51.85 | 42.23 | 43.51 | 48.36
  Smoking (Unknown) | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality.
  Alcohol consumption (drinker) | 64.29 | 62.72 | 62.21 | 64.25 | 59.83 | 58.20
  Alcohol consumption (non-drinker) | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 12.14 | 15.47 | 13.16 | 15.48 | 13.11
  Alcohol consumption (ex-drinker) | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 21.68 | 17.05 | 14.87 | 17.36 | 22.95
  Alcohol consumption (Unknown) | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 3.47 | 5.27 | 7.72 | 7.32 | 5.74

14. Secondary Outcome: Baseline Characteristics (as Measured by Life Style Factors (BMI)) of Patients Starting Index Prescriptions Off-label
Description: Baseline characteristics of patients (as measured by life style factors (BMI)) who initiated index prescriptions (empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists)) off-label is presented. Use of empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs in other types of diabetes (other than T2DM) or without diabetes or in people younger than 18 years old or in women during pregnancy or during breastfeeding is considered as off-label. As per CPRD guideline, no cell that contains <5 events should be reported to protect patient confidentiality. Since empagliflozin group reported <5 events for all off-label categories except for unspecified DM therefore baseline characteristics are presented for only unspecified DM category.
Time Frame: Baseline
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Kilogram per square meter (kg/m2)
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Number analyzed (Participants) | 14 | 336 | 536 | 808 | 427 | 120
Kilogram per square meter (kg/m2) | 33.29 (5.77) | 34.71 (6.66) | 31.73 (6.40) | 32.40 (7.21) | 30.81 (6.49) | 36.50 (6.43)

15. Secondary Outcome: Baseline Characteristics (as Measured by Life Style Factors (Blood Pressure)) of Patients Starting Index Prescriptions Off-label
Description: Baseline characteristics of patients (as measured by life style factors (blood pressure)) who initiated index prescriptions (empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists)) off-label is presented. Use of empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs in other types of diabetes (other than T2DM) or without diabetes or in people younger than 18 years old or in women during pregnancy or during breastfeeding is considered as off-label. As per CPRD guideline, no cell that contains <5 events should be reported to protect patient confidentiality. Since empagliflozin group reported <5 events for all off-label categories except for unspecified DM therefore baseline characteristics are presented for only unspecified DM category.
Time Frame: Baseline
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Number analyzed (Participants) | 14 | 346 | 569 | 1049 | 478 | 122
Millimeter of mercury (mmHg)
  SBP: number analyzed (Participants) | 14 | 309 | 519 | 782 | 413 | 108
  SBP | 131.43 (12.79) | 133.94 (15.97) | 134.41 (16.19) | 134.95 (16.96) | 130.86 (14.86) | 133.18 (14.58)
  DBP: number analyzed (Participants) | 14 | 308 | 517 | 786 | 414 | 108
  DBP | 75.43 (5.24) | 76.85 (9.93) | 75.42 (9.66) | 78.74 (11.02) | 75.89 (10.00) | 75.97 (10.20)

16. Secondary Outcome: Baseline Characteristics (as Measured b Yglycated Haemoglobin (HbA1c)) of Patients Starting Index Prescriptions Off-label
Description: Baseline characteristics of patients (as measured by glycated haemoglobin (HbA1c)) who initiated index prescriptions (empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists)) off-label is presented. Use of empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs in other types of diabetes (other than T2DM) or without diabetes or in people younger than 18 years old or in women during pregnancy or during breastfeeding is considered as off-label. As per CPRD guideline, no cell that contains <5 events should be reported to protect patient confidentiality. Since empagliflozin group reported <5 events for all off-label categories except for unspecified DM therefore baseline characteristics are presented for only unspecified DM category.
Time Frame: Baseline
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimole per mole (mmol/mol)
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Number analyzed (Participants) | 13 | 290 | 497 | 722 | 371 | 105
Millimole per mole (mmol/mol) | 79.69 (13.79) | 82.17 (18.45) | 74.70 (17.55) | 72.29 (23.94) | 79.21 (23.55) | 83.23 (19.86)

17. Secondary Outcome: Baseline Characteristics (as Measured by Laboratory Tests) of Patients Starting Index Prescriptions Off-label
Description: Baseline characteristics of patients (as measured by laboratory tests) who initiated index prescriptions (empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists)) off-label are presented. Use of empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs in other types of diabetes (other than T2DM) or without diabetes or in people younger than 18 years old or in women during pregnancy or during breastfeeding is considered as off-label. As per CPRD guideline, no cell that contains <5 events should be reported to protect patient confidentiality. Since empagliflozin group reported <5 events for all off-label categories except for unspecified DM therefore baseline characteristics are presented for only unspecified DM category.
Time Frame: Baseline
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimole per liter (mmol/L)
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Number analyzed (Participants) | 14 | 346 | 569 | 1049 | 478 | 122
Millimole per liter (mmol/L)
  TC: number analyzed (Participants) | 13 | 325 | 523 | 782 | 401 | 111
  TC | 3.96 (0.93) | 4.33 (1.14) | 4.25 (1.18) | 4.95 (1.29) | 4.49 (1.24) | 4.40 (1.17)
  HDL: number analyzed (Participants) | 13 | 289 | 466 | 722 | 370 | 100
  HDL | 1.16 (0.39) | 1.14 (0.32) | 1.17 (0.31) | 1.22 (0.39) | 1.19 (0.31) | 1.15 (0.35)
  LDL: number analyzed (Participants) | 8 | 241 | 378 | 576 | 288 | 79
  LDL | 2.08 (1.05) | 2.24 (0.96) | 2.15 (0.86) | 2.73 (1.02) | 2.27 (0.95) | 2.09 (0.98)
  TG: number analyzed (Participants) | 9 | 269 | 426 | 650 | 322 | 97
  TG | 1.84 (1.17) | 2.38 (1.76) | 2.15 (1.47) | 2.43 (2.34) | 2.27 (1.51) | 2.38 (1.41)

18. Secondary Outcome: Baseline Characteristics (as Measured by Estimated Glomerular Filtration Rate (eGFR)) of Patients Starting Index Prescriptions Off-label
Description: Baseline characteristics of patients (as measured by estimated glomerular filtration rate (eGFR)) who initiated index prescriptions (empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists)) off-label is presented. Use of empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs in other types of diabetes (other than T2DM) or without diabetes or in people younger than 18 years old or in women during pregnancy or during breastfeeding is considered as off-label. As per CPRD guideline, no cell that contains <5 events should be reported to protect patient confidentiality. Since empagliflozin group reported <5 events for all off-label categories except for unspecified DM therefore baseline characteristics are presented for only unspecified DM category.
Time Frame: Baseline
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Milliliters per minute (ml/min)
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Number analyzed (Participants) | 14 | 330 | 550 | 887 | 435 | 119
Milliliters per minute (ml/min) | 91.05 (17.01) | 93.23 (16.89) | 78.52 (25.20) | 89.36 (20.99) | 82.31 (25.09) | 85.57 (21.19)

19. Secondary Outcome: Baseline Characteristics (as Measured by Creatinine Serum (SCR)) of Patients Starting Index Prescriptions Off-label
Description: Baseline characteristics of patients (as measured by creatinine serum (SCR)) who initiated index prescriptions (empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists)) off-label is presented. Use of empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs in other types of diabetes (other than T2DM) or without diabetes or in people younger than 18 years old or in women during pregnancy or during breastfeeding is considered as off-label. As per CPRD guideline, no cell that contains <5 events should be reported to protect patient confidentiality. Since empagliflozin group reported <5 events for all off-label categories except for unspecified DM therefore baseline characteristics are presented for only unspecified DM category.
Time Frame: Baseline
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Number analyzed (Participants) | 14 | 330 | 550 | 887 | 435 | 119
Micromoles per liter (umol/L) | 74.21 (17.76) | 74.10 (19.28) | 92.89 (47.49) | 78.21 (23.53) | 87.41 (43.47) | 81.97 (26.08)

20. Secondary Outcome: Baseline Characteristics (as Measured by Comorbidities) of Patients Starting Index Prescriptions Off-label
Description: Baseline characteristics of patients (as measured by comorbidities) who initiated index prescriptions (empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists)) off-label are presented. Use of empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs in other types of diabetes (other than T2DM) or without diabetes or in people younger than 18 years old or in women during pregnancy or during breastfeeding is considered as off-label. As per CPRD guideline, no cell that contains <5 events should be reported to protect patient confidentiality. Since empagliflozin group reported <5 events for all off-label categories except for unspecified DM therefore baseline characteristics are presented for only unspecified DM category.
Time Frame: Baseline
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Number analyzed (Participants) | 14 | 346 | 569 | 1049 | 478 | 122
Percentage of Participants
  Diabetes complications | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 47.69 | 37.26 | 14.59 | 27.41 | 40.98
  Thyroid disorders | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 5.20 | 6.33 | 8.29 | 5.44 | 4.92
  Cancer | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 2.89 | 5.98 | 4.96 | 6.90 | 5.74
  Cardiovascular disorders | 35.71 | 44.51 | 51.67 | 41.37 | 44.98 | 43.44
  Infections | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 2.02 | 2.99 | 3.91 | 3.56 | 4.10
  Kidney disease | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 8.96 | 23.90 | 9.34 | 15.06 | 15.57
  Polycystic Ovary Syndrome (PCO), females only | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 11.70 | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality.
  Obesity | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 24.57 | 15.29 | 17.16 | 13.81 | 27.87
  Respiratory | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 15.90 | 18.63 | 16.02 | 18.41 | 22.13
  Pancreatitis | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 0.95 | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality.
  Bone disorders | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 8.67 | 9.31 | 10.96 | 11.30 | 4.92

21. Secondary Outcome: Baseline Characteristics (as Measured by Concomitant Medications) of Patients Starting Index Prescriptions Off-label
Description: Baseline characteristics of patients (as measured by concomitant medications) who initiated index prescriptions (empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs (comprising DPP-4i, metformin, SU and GLP-1 agonists)) off-label are presented. Use of empagliflozin, other SGLT-2i or other commonly used non-insulin GLDs in other types of diabetes (other than T2DM) or without diabetes or in people younger than 18 years old or in women during pregnancy or during breastfeeding is considered as off-label. As per CPRD guideline, no cell that contains <5 events should be reported to protect patient confidentiality. Since empagliflozin group reported <5 events for all off-label categories except for unspecified DM therefore baseline characteristics are presented for only unspecified DM category. Subjects taking medication up to 60 days before index date are presented.
Time Frame: Baseline
Population: as for outcome 12
Measure: Number; unit: Percentage of Participants
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Number analyzed (Participants) | 14 | 346 | 569 | 1049 | 478 | 122
Percentage of Participants
  Insulin | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 33.82 | 12.13 | 9.25 | 3.77 | 36.07
  Non-insulin GLDs | 85.71 | 91.33 | 85.06 | 11.44 | 70.08 | 84.43
  Cardiovascular medications | 85.71 | 77.17 | 79.96 | 52.24 | 66.53 | 74.59
  Lipid-regulating Drugs | 85.71 | 75.14 | 75.22 | 38.42 | 58.58 | 72.95
  Oral Corticosteroids | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 1.45 | 3.16 | 4.29 | 3.56 | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality.
  Non-steroidal anti-inflammatory drugs | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 10.12 | 6.85 | 8.87 | 8.79 | 13.93
  Psycholeptics | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 8.09 | 5.98 | 7.15 | 8.79 | 5.74
  Antipsychotics | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 3.76 | 3.87 | 3.43 | 2.72 | 4.92
  Antidepressants | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 30.92 | 26.01 | 21.83 | 26.99 | 32.79
  Opiates | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 28.61 | 22.14 | 19.73 | 22.38 | 26.23
  Anti-Epilepsy, Anticonvulsants | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 15.90 | 10.02 | 9.44 | 6.90 | 13.11
  Anti-Parkinson, Dopamine agonists | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 2.31 | 2.64 | 2.29 | 2.93 | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality.
  Agents for dementia | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 1.05 | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality. | 1.26 | NA — CPRD policy is that no cell that contains <5 events should be reported, to protect patient confidentiality.

ADVERSE EVENTS:
Description: Based on current guidelines from the International Society for Pharmacoepidemiology and good pharmacovigilance practices (GVP) Module VI, reporting of adverse reactions in noninterventional studies conducted using electronic claims and health care records (based on use of secondary data) is not required.
Arm/Group | Empagliflozin | Other SGLT-2i | Dipeptidyl Peptidase-4 Inhibitors (DPP-4i) | Metformin | Sulfonylureas (SU) | Glucagon-like Peptide-1 (GLP-1) Agonists
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The utilization of empagliflozin in the first year after launch was not as high as other exposure categories.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.